CLINICAL TRIAL: NCT02418026
Title: Improving Cesarean Section Experience Through Hypnotherapy: a Prospective Single Center Case-control Study
Brief Title: Improving Cesarean Section Experience Through Hypnotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Rochelle Ré Aunis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014/P01/034
Record Dates: First submitted 2015-04-07; First posted 2015-04-16 (Estimated); Results first posted 2017-03-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cesarean Section; Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): women who attended the obstetrics department for a scheduled or unplanned cesarean section and who benefited from general care
- Hypnosis (Experimental): women who attended the obstetrics department for a scheduled or unplanned cesarean section and who benefited from a hypnosis session during the surgery in addition to general care
  Interventions: Other: hypnosis

INTERVENTIONS:
Other: hypnosis — Conversational hypnotic induction and therapeutic suggestions
  Arms: Hypnosis

SUMMARY:
Cesarean section rates continue to increase worldwide, particularly in middle- and high-income countries. In France, the rate has now stabilized around 20 %. Cesarean section is a particular way of giving birth, sometimes desired, but sometimes feared. If some women do not feel affected by this way of giving birth, it is more difficult for others to live with. In this way, not being able to give birth trough natural way may be disturbing in motherhood. At La Rochelle hospital, more than 230 healthcare providers have been trained according to Erickson's hypnosis methodology. Among them, 40 are part of the anesthesia department and a committee oversees the hypnotherapist activities in pain management. The objective of the present study is to assess the benefit of hypnosis session for improving experience and reducing anxiety in women giving birth through surgery.

DETAILED DESCRIPTION:
Nonpharmacological approaches for pain management, either as a primary method or as a complement to pharmacological approaches, are suggested for a better perinatal management. The investigators assessed the use of conversational hypnotic induction and therapeutic suggestions during cesarean section as a complement to pharmacological strategy. Women giving birth through scheduled or unplanned cesarean section and who accepted hypnotherapy session were compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* scheduled or unplanned cesarean section
* Informed consent

Exclusion Criteria:

* Refusal of the patient to participate in the study
* Not French speaking
* Patients under guardianship

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2013-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine DELAVAUX, Principal Investigator — Groupe Hospitalier de la Rochelle Ré Aunis

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Hypnosis
Started | 44 | 35
Completed | 44 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Hypnosis | Total
Number analyzed (Participants) | 44 | 35 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (5.7) | 31.2 (5.3) | 30.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 35 | 79
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 44 | 35 | 79

OUTCOME MEASURES:

1. Primary Outcome: Wellbeing Measured Using a Comfort Scale
Description: The comfort scale is a numeric rating scale ranging from 0 to 10 : 0 corresponds to "no comfort" and 10 corresponds to "most comfortable".
Time Frame: just after surgery, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
units on a scale | 6.7 (1.7) | 8.0 (1.4)

2. Secondary Outcome: Wellbeing Measured Using a Comfort Scale
Description: as for outcome 1
Time Frame: Day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
units on a scale | 7.8 (1.5) | 8.0 (1.5)

3. Secondary Outcome: Wellbeing Measured Using a Comfort Scale
Description: as for outcome 1
Time Frame: Day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
units on a scale | 8.9 (1.4) | 8.8 (1.2)

4. Secondary Outcome: Score at Numeric Pain Rating Scale
Description: The numeric pain rating scale ranges from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: just after surgery, up to 1 hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
units on a scale | 2.0 (1.9) | 1.3 (1.4)

5. Secondary Outcome: Score at Numeric Pain Rating Scale
Description: The numeric pain rating scale ranges from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: day 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
units on a scale | 2.1 (1.4) | 2.1 (1.1)

6. Secondary Outcome: Score at Numeric Pain Rating Scale
Description: The numeric pain rating scale range from 0 (no pain) to 10 (worst pain imaginable)
Time Frame: day 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
units on a scale | 1.1 (1.6) | 1.1 (1.1)

7. Secondary Outcome: Mean Blood Pressure
Time Frame: preoperative, up to 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
mm Hg | 96 (11) | 101 (14)

8. Secondary Outcome: Mean Blood Pressure
Time Frame: during surgery (average), up to 2 hours
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
mm Hg | 85 (10) | 84 (10)

9. Secondary Outcome: Mean Blood Pressure
Time Frame: for 2 hours in the recovery room at regular intervals (average)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
mm Hg | 87 (10) | 88 (10)

10. Secondary Outcome: Mean Pulse
Time Frame: preoperative, up to 2 hours
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
bpm | 95 (17) | 94 (17)

11. Secondary Outcome: Mean Pulse
Time Frame: during surgery (average), up to 2 hours
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
bpm | 90 (13) | 90 (15)

12. Secondary Outcome: Mean Pulse
Time Frame: for 2 hours in the recovery room at regular intervals (average)
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
bpm | 86 (15) | 84 (13)

13. Secondary Outcome: Non-steroidal Anti-inflammatory Drug Intake
Time Frame: day 3
Measure: Number; unit: participants
Arm/Group | Control | Hypnosis
Number analyzed (Participants) | 44 | 35
participants | 43 | 18

ADVERSE EVENTS:
Arm/Group | Control | Hypnosis
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/35
Other Adverse Events (participants affected / at risk) | 0/44 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes